CLINICAL TRIAL: NCT01948986
Title: A Phase 1, Non-Randomized, Open-Label, Single Dose Study to Evaluate the Effect of Renal Impairment on the Pharmacokinetics, Pharmacodynamics, Safety and Tolerability of Ertugliflozin in Subjects With Type 2 Diabetes Mellitus
Brief Title: Effect of Renal Impairment on the Pharmacokinetics, Pharmacodynamics, Safety and Tolerability of Ertugliflozin in Participants With Type 2 Diabetes Mellitus (MK-8835-009)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 8835-009; B1521023 (Other: Pfizer protocol number); MK-8835-009 (Other: Merck protocol number)
Record Dates: First submitted 2013-09-20; First posted 2013-09-24 (Estimated); Results first posted 2019-02-18 (Actual); Last update posted 2019-02-18 (Actual); Status verified 2018-10

CONDITIONS: Renal Impairment; Type 2 Diabetes Mellitus
MeSH Terms: conditions — Renal Insufficiency; Diabetes Mellitus, Type 2 | interventions — ertugliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Ertugliflozin 15 mg (T2DM with Normal Renal Function) (Experimental): Ertugliflozin (15 mg), oral, administered in participants with T2DM and with normal renal function
  Interventions: Drug: Ertugliflozin
- Ertugliflozin 15 mg (T2DM with Mild Renal Impairment) (Experimental): Ertugliflozin (15 mg), oral, administered in participants with T2DM and with mild renal impairment
  Interventions: Drug: Ertugliflozin
- Ertugliflozin 15 mg (T2DM with Moderate Renal Impairment) (Experimental): Ertugliflozin (15 mg), oral, administered in participants with T2DM and with moderate renal impairment
  Interventions: Drug: Ertugliflozin
- Ertugliflozin 15 mg (T2DM with Severe Renal Impairment) (Experimental): Ertugliflozin (15 mg), oral, administered in participants with T2DM and with severe renal impairment
  Interventions: Drug: Ertugliflozin
- Ertugliflozin, 15 mg (Healthy Part. with Normal Renal Funct.) (Experimental): Ertugliflozin (15 mg), oral, administered in participants with healthy participants and with normal renal function
  Interventions: Drug: Ertugliflozin

INTERVENTIONS:
Drug: Ertugliflozin — Single oral administration of 3 X 5 mg tablets.
  Other Names: MK-8835

SUMMARY:
This is a study to evaluate the effect of renal impairment on the pharmacokinetics, pharmacodynamics, safety and tolerability of ertugliflozin in participants with type 2 diabetes mellitus (T2DM) and in healthy participants with normal renal function.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) of approximately 18 to 40 kg/m^2
* Stable renal function
* Male or female not of reproductive potential
* Female of reproductive potential must agree or have their partner agree to use 2 acceptable methods of contraception
* Healthy subjects determined to be healthy by investigator screening
* T2DM participants have a diagnosis of T2DM as per American Diabetes Association guidelines
* T2DM participants to be on a stable anti-hyperglycemic regimen with no new drug or drug dosage within 8 weeks of study participation. Variations in daily dose of insulin up to 10% are permitted.

Exclusion Criteria:

* A positive urine drug screen for drugs of abuse or recreational drugs
* Pregnant or nursing females
* History of abuse of alcohol or illicit drugs
* Significant renal or urinary disease within 6 months of study participation
* History of malignancy within the past 5 years basal cell carcinoma of the skin or cervical cancer in situ
* History of human immunodeficiency virus (HIV)
* History of blood dyscrasias or any disorders causing hemolysis or unstable red blood cells
* Any acute disease state (eg, , vomiting, fever, diarrhea) within 7 days before study participation
* Treatment with an investigational drug within 30 days of study participation
* Use of herbal supplements within 28 days prior to study participation
* Any clinically significant malabsorption condition
* Blood donation (excluding plasma donations) of approximately 1 pint within 56 days prior to study participation
* History of sensitivity to ertugliflozin or other Sodium-Glucose co-Transporter 2 (SGLT2) inhibitors
* History of sensitivity to heparin or heparin-induced thrombocytopenia
* Unwilling or unable to comply with the study Lifestyle Guidelines
* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease including clinically relevant and significant drug allergies
* Use of prescription drugs (hormonal methods of birth control are allowed), vitamins and dietary supplements within 7 days of study participation
* For T2DM participants, history of type 1 diabetes mellitus or a history of ketoacidosis
* For T2DM participants, clinically significant electrocardiogram abnormality
* For T2DM participants, history of myocardial infarction, unstable angina, coronary revascularization, stroke or transient ischemic attack within 3 months of study participation
* For T2DM participants, heart failure defined as New York Heart Association Functional Class III-IV
* For T2DM participants, renal allograft recipients
* For T2DM participants, requiring dialysis
* For T2DM participants, strict fluid restriction
* For T2DM participants, urinary incontinence
* For T2DM participants, acute renal disease
* For T2DM participants, significant hepatic, cardiac, or pulmonary disease or clinically nephrotic
* For T2DM participants, prescription and over-the-counter medication that is not taken according to a stable regimen for 7 days before study participation
* For T2DM participants, on metformin should not be enrolled if their baseline renal function is outside the approved product labeling
* For T2DM participants receiving any of the following medications within 7 days of study participation: 1. Other SGLT2 inhibitors (eg, dapagliflozin, canagliflozin, empagliflozin); 2. Other injectable anti-hyperglycemic agents including pramlintide or Glucagon-like peptide-1 (GLP-1) analogues; 3. Any immunosuppressive drugs, including cyclosporine, tacrolimus, sirolimus; 4. Oral corticosteroids (note that inhaled, nasal and topical corticosteroids are permitted); 5. Any potent drug-metabolizing enzyme-inducing drug, including rifampin, phenytoin, and carbamazepine; 6. Probenecid, valproic acid, gemfibrozil.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2013-10-01 (Actual); Primary Completion 2014-10-06 (Actual); Study Completion 2014-10-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Sahasrabudhe V, Terra SG, Hickman A, Saur D, Shi H, O'Gorman M, Zhou Z, Cutler DL. The Effect of Renal Impairment on the Pharmacokinetics and Pharmacodynamics of Ertugliflozin in Subjects With Type 2 Diabetes Mellitus. J Clin Pharmacol. 2017 Nov;57(11):1432-1443. doi: 10.1002/jcph.955. Epub 2017 Jul 13. PMID 28703316
- [Derived] Fediuk DJ, Sahasrabudhe V, Dawra VK, Zhou S, Sweeney K. Population Pharmacokinetic Analyses of Ertugliflozin in Select Ethnic Populations. Clin Pharmacol Drug Dev. 2021 Nov;10(11):1297-1306. doi: 10.1002/cpdd.970. Epub 2021 Jul 2. PMID 34213819
- [Derived] Marshall JC, Liang Y, Sahasrabudhe V, Tensfeldt T, Fediuk DJ, Zhou S, Krishna R, Dawra VK, Wood LS, Sweeney K. Meta-Analysis of Noncompartmental Pharmacokinetic Parameters of Ertugliflozin to Evaluate Dose Proportionality and UGT1A9 Polymorphism Effect on Exposure. J Clin Pharmacol. 2021 Sep;61(9):1220-1231. doi: 10.1002/jcph.1866. Epub 2021 Jun 19. PMID 33813736

RESULTS

PARTICIPANT FLOW:
Groups:
- Ertugliflozin 15 mg (T2DM With Normal Renal Function): Ertugliflozin (15 mg), oral, administered in participants with Type 2 Diabetes Mellitus (T2DM) and with normal renal function
- Ertugliflozin 15 mg (T2DM and With Severe Renal Impairment): Ertugliflozin (15 mg), oral, administered in participants with T2DM and with severe renal impairment
- Ertugliflozin 15 mg (Healthy Part. With Normal Renal Function): Ertugliflozin (15 mg), oral, administered in participants with healthy participants and with normal renal function
Period: Overall Study
Arm/Group | Ertugliflozin 15 mg (T2DM With Normal Renal Function) | Ertugliflozin 15 mg (T2DM With Mild Renal Impairment) | Ertugliflozin 15 mg (T2DM With Moderate Renal Impairment) | Ertugliflozin 15 mg (T2DM and With Severe Renal Impairment) | Ertugliflozin 15 mg (Healthy Part. With Normal Renal Function)
Started | 6 | 8 | 8 | 6 | 8
Completed | 6 | 8 | 8 | 6 | 8
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Renal function groups were based on body surface area (BSA)-unnormalized estimated glomerular filtration rate (eGFR).
Groups:
- Total: Total of all reporting groups
Arm/Group | Ertugliflozin 15 mg (T2DM With Normal Renal Function) | Ertugliflozin 15 mg (T2DM With Mild Renal Impairment) | Ertugliflozin 15 mg (T2DM With Moderate Renal Impairment) | Ertugliflozin 15 mg (T2DM and With Severe Renal Impairment) | Ertugliflozin 15 mg (Healthy Part. With Normal Renal Function) | Total
Number analyzed (Participants) | 6 | 8 | 8 | 6 | 8 | 36
Age, Continuous [Mean (Full Range); unit: Years] | 63.2 (3.5) [60 to 68] | 66.4 (2.4) [63 to 70] | 65.8 (7.9) [54 to 76] | 61.2 (10.3) [49 to 76] | 64.3 (3.9) [60 to 70] | 64.4 [60 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 5 | 4 | 0 | 3 | 13
  Male | 5 | 3 | 4 | 6 | 5 | 23
Baseline Urinary Glucose Excretion (UGE) [Median (Full Range); unit: Grams] — Participants were asked to void at the end of each prescribed interval with forced voids prior to start and at the end of each interval.
  Grams | 8.2 (10.49) [0.1 to 29.0] | 0.1 (10.21) [0.0 to 29.0] | 0.2 (0.93) [0.0 to 2.7] | 2.3 (3.44) [0.1 to 8.9] | 0.1 (0.04) [0.0 to 0.1] | 1.8 [0.0 to 29.0]
Baseline eGFR [Mean (Full Range); unit: mL/min/1.73 m²] — Mean of screening BSA-normalized eGFR which was the average of the 2 screening eGFR values that were based on serum creatinine values obtained on 2 occasions separated by at least 72 hours to 14 days.
  mL/min/1.73 m² | 92.1 (14.10) [79.1 to 115.0] | 64.7 (7.52) [55.5 to 78.0] | 37.1 (6.92) [25.9 to 43.7] | 17.0 (7.51) [6.8 to 25.7] | 88.5 (11.64) [74.3 to 103.1] | 60.5 [6.8 to 115.0]
Baseline Inhibition of Glucose Readsorption [Median (Full Range); unit: Percentage] — Inhibition of Glucose Reabsorption = 100 * UGE / ( eGFR(ML/MIN) * Weighted Mean Plasma Glucose * 0.0144). 0.0144 is a unit conversion factor used to make the ratio unitless.
  Percentage | 2.7 (3.45) [0.0 to 9.6] | 0.1 (5.17) [0.0 to 14.7] | 0.3 (1.05) [0.0 to 3.1] | 3.3 (19.42) [0.2 to 50.4] | 0.0 (0.02) [0.0 to 0.1] | 1.1 [0.0 to 50.4]
Baseline Fluid Balance [Median (Full Range); unit: Milliliters] — Fluid balance = fluid intake - urine output. Fluid intake was measured during interval of -48 to -24 hours prior to dosing at Baseline.
  Milliliters | -644.0 (668.11) [-1355.0 to 635.0] | -274.8 (570.44) [-920.0 to 702.0] | 238.8 (763.10) [-963.0 to 1055.0] | -267.5 (430.85) [-830.0 to 320] | -359.5 (693.65) [-1780.0 to 164.0] | -243.1 [-1780.0 to 1055.0]

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration-Time Profile for Ertugliflozin From Time 0 Extrapolated to Infinite Time (AUCinf)
Description: Area under the plasma concentration-time profile from Time 0 extrapolated to infinite time. Blood samples were taken at pre-dose up to 96 hours post-dose, from which the concentration of ertugliflozin was determined. Geometric Coefficient of Variation was reported as a percent.
Time Frame: Time 0 (predose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, and 96 hours post-dose
Population: The analysis population was defined as all treated participants who had at least one concentration measurement for AUCinf.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng•hr/mL
Arm/Group | Ertugliflozin 15 mg (T2DM With Normal Renal Function) | Ertugliflozin 15 mg (T2DM With Mild Renal Impairment) | Ertugliflozin 15 mg (T2DM With Moderate Renal Impairment) | Ertugliflozin 15 mg (T2DM and With Severe Renal Impairment) | Ertugliflozin 15 mg (Healthy Part. With Normal Renal Function)
Number analyzed (Participants) | 6 | 8 | 8 | 6 | 8
ng•hr/mL | 1199 (42) | 1908 (28) | 2075 (19) | 1895 (23) | 1236 (27)
Statistical Analysis 1: Comparison: Ertugliflozin 15 mg (T2DM With Normal Renal Function) vs Ertugliflozin 15 mg (Healthy Part. With Normal Renal Function); Test type: Superiority or Other; Ratio (Heathy Normal/T2DM Normal) = 103.07, 90% CI 2-sided [80.32 to 132.27] — The model was an ANOVA model with renal function group as a fixed effect. The ratios (and 90% CIs) are expressed as percentages
Statistical Analysis 2: Comparison: Ertugliflozin 15 mg (T2DM With Mild Renal Impairment) vs Ertugliflozin 15 mg (Healthy Part. With Normal Renal Function); Test type: Superiority or Other; Ratio (Mild Renal Impair./Pooled Norm.) = 156.34, 90% CI 2-sided [127.83 to 191.23] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Ertugliflozin 15 mg (T2DM With Moderate Renal Impairment) vs Ertugliflozin 15 mg (Healthy Part. With Normal Renal Function); Test type: Superiority or Other; Ratio (Mod. Renal Impair./Pooled Norm.) = 170.04, 90% CI 2-sided [139.02 to 207.98] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Ertugliflozin 15 mg (T2DM and With Severe Renal Impairment) vs Ertugliflozin 15 mg (Healthy Part. With Normal Renal Function); Test type: Superiority or Other; Ratio (Severe Renal Impair./Pooled Norm. = 155.26, 90% CI 2-sided [124.38 to 193.80] — [estimate comment as in outcome 1, analysis 1]

2. Primary Outcome: Area Under the Plasma Concentration-Time Profile for Ertugliflozin From Time 0 to the Time of the Last Quantifiable Concentration (AUClast)
Description: Area under the plasma concentration-time profile from Time 0 to the time of the last quantifiable concentration (Clast). Blood samples were taken at pre-dose up to 96 hours post-dose, from which the concentration of ertugliflozin was determined. Geometric Coefficient of Variation was reported as a percent.
Time Frame: Time 0 (predose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, and 96 hours post-dose
Population: The analysis population was defined as all treated participants who had at least one concentration measurement for AUClast.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng•hr/mL
Arm/Group | Ertugliflozin 15 mg (T2DM With Normal Renal Function) | Ertugliflozin 15 mg (T2DM With Mild Renal Impairment) | Ertugliflozin 15 mg (T2DM With Moderate Renal Impairment) | Ertugliflozin 15 mg (T2DM and With Severe Renal Impairment) | Ertugliflozin 15 mg (Healthy Part. With Normal Renal Function)
Number analyzed (Participants) | 6 | 8 | 8 | 6 | 8
ng•hr/mL | 1174 (42) | 1814 (27) | 2011 (18) | 1816 (23) | 1214 (27)
Statistical Analysis 1: Comparison: Ertugliflozin 15 mg (T2DM With Normal Renal Function) vs Ertugliflozin 15 mg (Healthy Part. With Normal Renal Function); Test type: Superiority or Other; Ratio (Heathy Normal/T2DM Normal) = 103.42, 90% CI 2-sided [80.66 to 132.61] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Ertugliflozin 15 mg (T2DM With Mild Renal Impairment) vs Ertugliflozin 15 mg (Healthy Part. With Normal Renal Function); Test type: Superiority or Other; Ratio (Mild Renal Impair./Pooled Norm.) = 151.63, 90% CI 2-sided [124.05 to 185.34] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Ertugliflozin 15 mg (T2DM With Moderate Renal Impairment) vs Ertugliflozin 15 mg (Healthy Part. With Normal Renal Function); Test type: Superiority or Other; Ratio (Mod. Renal Impair./Pooled Norm.) = 168.11, 90% CI 2-sided [137.53 to 205.49] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Ertugliflozin 15 mg (T2DM and With Severe Renal Impairment) vs Ertugliflozin 15 mg (Healthy Part. With Normal Renal Function); Test type: Superiority or Other; Ratio (Severe Renal Impair./Pooled Norm. = 151.80, 90% CI 2-sided [121.69 to 189.36] — [estimate comment as in outcome 1, analysis 1]

3. Primary Outcome: Apparent Clearance (CL/F) for Plasma Ertugliflozin
Description: CL/F is a calculation of the rate at which a drug is removed from the body via renal, hepatic and other clearance pathways, expressed as volume (milliliters) per unit of time (minutes). Blood samples were taken at pre-dose up to 96 hours post-dose, from which the concentration of ertugliflozin was determined. Geometric Coefficient of Variation was reported as a percent.
Time Frame: Time 0 (predose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, and 96 hours post-dose
Population: The analysis population was defined as all treated participants who had at least one concentration measurement for CL/F.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/min
Arm/Group | Ertugliflozin 15 mg (T2DM With Normal Renal Function) | Ertugliflozin 15 mg (T2DM With Mild Renal Impairment) | Ertugliflozin 15 mg (T2DM With Moderate Renal Impairment) | Ertugliflozin 15 mg (T2DM and With Severe Renal Impairment) | Ertugliflozin 15 mg (Healthy Part. With Normal Renal Function)
Number analyzed (Participants) | 6 | 8 | 8 | 6 | 8
mL/min | 208.8 (42) | 130.9 (28) | 120.4 (19) | 132.0 (23) | 202.1 (27)

4. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) for Ertugliflozin
Description: Cmax is a measure of the maximum amount of drug in the plasma after the dose is given. Blood samples were taken at pre-dose up to 96 hours post-dose, from which the concentration of ertugliflozin was determined. Geometric Coefficient of Variation was reported as a percent.
Time Frame: Time 0 (predose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, and 96 hours post-dose
Population: The analysis population was defined as all treated participants who had at least one concentration measurement for Cmax.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Ertugliflozin 15 mg (T2DM With Normal Renal Function) | Ertugliflozin 15 mg (T2DM With Mild Renal Impairment) | Ertugliflozin 15 mg (T2DM With Moderate Renal Impairment) | Ertugliflozin 15 mg (T2DM and With Severe Renal Impairment) | Ertugliflozin 15 mg (Healthy Part. With Normal Renal Function)
Number analyzed (Participants) | 6 | 8 | 8 | 6 | 8
ng/mL | 215.9 (35) | 313.1 (30) | 305.7 (23) | 196.4 (28) | 219.3 (26)
Statistical Analysis 1: Comparison: Ertugliflozin 15 mg (T2DM With Normal Renal Function) vs Ertugliflozin 15 mg (Healthy Part. With Normal Renal Function); Test type: Superiority or Other; Ratio (Heathy Normal/T2DM Normal) = 101.57, 90% CI 2-sided [78.83 to 130.87] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Ertugliflozin 15 mg (T2DM With Mild Renal Impairment) vs Ertugliflozin 15 mg (Healthy Part. With Normal Renal Function); Test type: Superiority or Other; Ratio (Mild Renal Impair./Pooled Norm.) = 143.74, 90% CI 2-sided [117.15 to 176.37] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Ertugliflozin 15 mg (T2DM With Moderate Renal Impairment) vs Ertugliflozin 15 mg (Healthy Part. With Normal Renal Function); Test type: Superiority or Other; Ratio (Mod. Renal Impair./Pooled Norm.) = 140.37, 90% CI 2-sided [114.40 to 172.23] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Ertugliflozin 15 mg (T2DM and With Severe Renal Impairment) vs Ertugliflozin 15 mg (Healthy Part. With Normal Renal Function); Test type: Superiority or Other; Ratio (Severe Renal Impair./Pooled Norm. = 90.18, 90% CI 2-sided [71.99 to 112.96] — [estimate comment as in outcome 1, analysis 1]

5. Primary Outcome: Time for Cmax (Tmax) for Plasma Ertugliflozin
Description: Tmax is a measure of the time to reach the maximum concentration in the plasma after the drug dose and is observed directly from data as time of first occurrence. Blood samples were taken at pre-dose up to 96 hours post-dose, from which the concentration of ertugliflozin was determined.
Time Frame: Time 0 (predose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, and 96 hours post-dose
Population: The analysis population was defined as all treated participants who had at least one concentration measurement for Tmax.
Measure: Median (Full Range); unit: Hours
Arm/Group | Ertugliflozin 15 mg (T2DM With Normal Renal Function) | Ertugliflozin 15 mg (T2DM With Mild Renal Impairment) | Ertugliflozin 15 mg (T2DM With Moderate Renal Impairment) | Ertugliflozin 15 mg (T2DM and With Severe Renal Impairment) | Ertugliflozin 15 mg (Healthy Part. With Normal Renal Function)
Number analyzed (Participants) | 6 | 8 | 8 | 6 | 8
Hours | 1.00 [1.00 to 1.50] | 1.50 [1.00 to 2.00] | 1.50 [0.500 to 2.00] | 1.51 [0.500 to 3.02] | 1.00 [1.00 to 2.00]

6. Primary Outcome: Terminal Half-Life (t1/2) for Plasma Ertugliflozin
Description: T1/2 is the time required for a given drug concentration in the plasma to decrease by 50%. T1/2 = Loge(2)/kel, where kel was the terminal phase rate constant calculated by a linear regression of the log-linear concentration-time curve. Blood samples were taken at pre-dose up to 96 hours post-dose, from which the concentration of ertugliflozin was determined.
Time Frame: Time 0 (predose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, and 96 hours post-dose
Population: The analysis population was defined as all treated participants who had at least one concentration measurement for t1/2.
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Ertugliflozin 15 mg (T2DM With Normal Renal Function) | Ertugliflozin 15 mg (T2DM With Mild Renal Impairment) | Ertugliflozin 15 mg (T2DM With Moderate Renal Impairment) | Ertugliflozin 15 mg (T2DM and With Severe Renal Impairment) | Ertugliflozin 15 mg (Healthy Part. With Normal Renal Function)
Number analyzed (Participants) | 6 | 8 | 8 | 6 | 8
Hours | 14.62 (6.37) | 25.94 (13.98) | 22.89 (7.35) | 24.17 (5.98) | 17.71 (3.53)

7. Primary Outcome: Apparent Volume of Distribution Following Oral Administration (Vz/F) for Plasma Ertugliflozin
Description: VzF is the apparent volume of distribution during terminal phase after oral / extravascular administration. VzF = Dose/(AUCinf × kel) where kel was the terminal phase rate constant calculated by a linear regression of the log-linear concentration-time curve. Blood samples were taken at pre-dose up to 96 hours post-dose, from which the concentration of ertugliflozin was determined. Geometric Coefficient of Variation was reported as a percent.
Time Frame: Time 0 (predose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, and 96 hours post-dose
Population: The analysis population was defined as all treated participants who had at least one concentration measurement for Vz/F.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | Ertugliflozin 15 mg (T2DM With Normal Renal Function) | Ertugliflozin 15 mg (T2DM With Mild Renal Impairment) | Ertugliflozin 15 mg (T2DM With Moderate Renal Impairment) | Ertugliflozin 15 mg (T2DM and With Severe Renal Impairment) | Ertugliflozin 15 mg (Healthy Part. With Normal Renal Function)
Number analyzed (Participants) | 6 | 8 | 8 | 6 | 8
Liters | 239.7 (53) | 254.5 (50) | 228.3 (27) | 268.8 (41) | 304.5 (39)

8. Primary Outcome: Unbound Fraction (Fu) for Plasma Ertugliflozin
Description: Fraction of unbound (not protein-bound) drug in plasma. Fu is determined using in vitro equilibrium dialysis method: concentration in buffer at equilibrium/concentration in plasma at equilibrium. Blood samples were taken at pre-dose up to 96 hours post-dose, from which the concentration of ertugliflozin was determined.
Time Frame: Time 0 (predose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, and 96 hours post-dose
Population: The analysis population was defined as all treated participants who had at least one concentration measurement for Fu.
Measure: Mean (Standard Deviation); unit: Percent of Unbound Drug
Arm/Group | Ertugliflozin 15 mg (T2DM With Normal Renal Function) | Ertugliflozin 15 mg (T2DM With Mild Renal Impairment) | Ertugliflozin 15 mg (T2DM With Moderate Renal Impairment) | Ertugliflozin 15 mg (T2DM and With Severe Renal Impairment) | Ertugliflozin 15 mg (Healthy Part. With Normal Renal Function)
Number analyzed (Participants) | 6 | 8 | 8 | 6 | 8
Percent of Unbound Drug | 0.03437 (0.0011219) | 0.03458 (0.0027696) | 0.03804 (0.0021287) | 0.04107 (0.0036621) | 0.03484 (0.0014822)

9. Primary Outcome: Cumulative Amount of Drug Recovered Unchanged in Urine to 96 Hours Post Dose (Ae96)
Description: Urine samples were taken at pre-dose up to 96 hours post-dose, from which the concentration of ertugliflozin was determined.
  Ae96 = Sum of [urine concentration × sample volume] for each collection interval from 0 to 96 hours post dose. Geometric Coefficient of Variation was reported as a percent.
Time Frame: 0-4, 4-8, 8-12, 12-24, 24-48, 48-72, and 72-96 hours after dosing on Day 1
Population: The analysis population was defined as all treated participants who had at least one concentration measurement for Ae96.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Milligrams
Arm/Group | Ertugliflozin 15 mg (T2DM With Normal Renal Function) | Ertugliflozin 15 mg (T2DM With Mild Renal Impairment) | Ertugliflozin 15 mg (T2DM With Moderate Renal Impairment) | Ertugliflozin 15 mg (T2DM and With Severe Renal Impairment) | Ertugliflozin 15 mg (Healthy Part. With Normal Renal Function)
Number analyzed (Participants) | 6 | 8 | 8 | 6 | 8
Milligrams | 0.1494 (55) | 0.1081 (54) | 0.09682 (21) | 0.05843 (40) | 0.1231 (48)

10. Primary Outcome: Percent of Dose Recovered Unchanged in Urine From 0 to 96 Hours Postdose (for Ertugliflozin Only) (Ae96%)
Description: Urine samples were taken at pre-dose up to 96 hours post-dose, from which the concentration of ertugliflozin was determined.
  Ae96% = Ae96 / Dose × 100 Ae96 = Sum of [urine concentration × sample volume] for each collection interval from 0 to 96 hours post dose. Geometric Coefficient of Variation was reported as a percent.
Time Frame: 0-4, 4-8, 8-12, 12-24, 24-48, 48-72, and 72-96 hours after dosing on Day 1
Population: The analysis population was defined as all treated participants who had at least one concentration measurement for Ae96.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percent
Arm/Group | Ertugliflozin 15 mg (T2DM With Normal Renal Function) | Ertugliflozin 15 mg (T2DM With Mild Renal Impairment) | Ertugliflozin 15 mg (T2DM With Moderate Renal Impairment) | Ertugliflozin 15 mg (T2DM and With Severe Renal Impairment) | Ertugliflozin 15 mg (Healthy Part. With Normal Renal Function)
Number analyzed (Participants) | 6 | 8 | 8 | 6 | 8
Percent | 0.9952 (55) | 0.7200 (54) | 0.6456 (21) | 0.3893 (40) | 0.8213 (48)

11. Primary Outcome: Renal Clearance (CLr) for Urinary Ertugliflozin
Description: Urine samples were taken at pre-dose up to 96 hours post-dose, from which the concentration of ertugliflozin was determined.
  CLr is Renal Clearance (Ae96 / AUC96), where Ae96 is the cumulative amount of drug recovered unchanged in urine to 96 hours post dose and AUC96 was the area under the concentration-time profile form time 0 to 96 hours. Geometric Coefficient of Variation was reported as a percent.
Time Frame: 0-4, 4-8, 8-12, 12-24, 24-48, 48-72, and 72-96 hours after dosing on Day 1
Population: The analysis population was defined as all treated participants who had at least one concentration measurement for CLr.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/min
Arm/Group | Ertugliflozin 15 mg (T2DM With Normal Renal Function) | Ertugliflozin 15 mg (T2DM With Mild Renal Impairment) | Ertugliflozin 15 mg (T2DM With Moderate Renal Impairment) | Ertugliflozin 15 mg (T2DM and With Severe Renal Impairment) | Ertugliflozin 15 mg (Healthy Part. With Normal Renal Function)
Number analyzed (Participants) | 6 | 8 | 8 | 6 | 8
mL/min | 2.092 (28) | 0.9872 (45) | 0.8024 (34) | 0.5360 (23) | 1.682 (33)
Statistical Analysis 1: Comparison: Ertugliflozin 15 mg (T2DM With Normal Renal Function) vs Ertugliflozin 15 mg (Healthy Part. With Normal Renal Function); Test type: Superiority or Other; Ratio (Heathy Normal/T2DM Normal) = 80.39, 90% CI 2-sided [59.41 to 108.76] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Ertugliflozin 15 mg (T2DM With Mild Renal Impairment) vs Ertugliflozin 15 mg (Healthy Part. With Normal Renal Function); Test type: Superiority or Other; Ratio (Mild Renal Impair./Pooled Norm.) = 53.46, 90% CI 2-sided [41.64 to 68.63] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Ertugliflozin 15 mg (T2DM With Moderate Renal Impairment) vs Ertugliflozin 15 mg (Healthy Part. With Normal Renal Function); Test type: Superiority or Other; Ratio (Mod. Renal Impair./Pooled Norm.) = 43.45, 90% CI 2-sided [33.85 to 55.78] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Ertugliflozin 15 mg (T2DM and With Severe Renal Impairment) vs Ertugliflozin 15 mg (Healthy Part. With Normal Renal Function); Test type: Superiority or Other; Ratio (Severe Renal Impair./Pooled Norm. = 29.02, 90% CI 2-sided [22.04 to 38.21] — [estimate comment as in outcome 1, analysis 1]

12. Primary Outcome: Number of Participants Who Experienced an Adverse Event (AE)
Description: An adverse event (AE) is defined as any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease associated with the use of a medical treatment or procedure, regardless of whether it is considered related to the medical treatment or procedure, that occurs during the course of the study.
Time Frame: Up to 19 days
Population: The analysis population was defined as all treated participants.
Measure: Number; unit: Participants
Arm/Group | Ertugliflozin 15 mg (T2DM With Normal Renal Function) | Ertugliflozin 15 mg (T2DM With Mild Renal Impairment) | Ertugliflozin 15 mg (T2DM With Moderate Renal Impairment) | Ertugliflozin 15 mg (T2DM and With Severe Renal Impairment) | Ertugliflozin 15 mg (Healthy Part. With Normal Renal Function)
Number analyzed (Participants) | 6 | 8 | 8 | 6 | 8
Participants | 1 | 2 | 2 | 3 | 4

13. Primary Outcome: Number of Participants Who Discontinued Study Due to an AE
Description: as for outcome 12
Time Frame: Up to 5 days
Population: The analysis population was defined as all treated participants.
Measure: Number; unit: Participants
Arm/Group | Ertugliflozin 15 mg (T2DM With Normal Renal Function) | Ertugliflozin 15 mg (T2DM With Mild Renal Impairment) | Ertugliflozin 15 mg (T2DM With Moderate Renal Impairment) | Ertugliflozin 15 mg (T2DM and With Severe Renal Impairment) | Ertugliflozin 15 mg (Healthy Part. With Normal Renal Function)
Number analyzed (Participants) | 6 | 8 | 8 | 6 | 8
Participants | 0 | 0 | 0 | 0 | 0

14. Primary Outcome: Area Under the Plasma Concentration-Time Profile for Glucuronide Metabolite PF-06481944 From Time 0 Extrapolated to Infinite Time (AUCinf)
Description: Area under the plasma concentration-time profile from Time 0 extrapolated to infinite time. Blood samples were taken at pre-dose up to 96 hours post-dose, from which the concentration of glucuronide metabolite PF 06481944 was determined. Geometric Coefficient of Variation was reported as a percent.
Time Frame: Time 0 (predose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, and 96 hours post-dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng•hr/mL
Arm/Group | Ertugliflozin 15 mg (T2DM With Normal Renal Function) | Ertugliflozin 15 mg (T2DM With Mild Renal Impairment) | Ertugliflozin 15 mg (T2DM With Moderate Renal Impairment) | Ertugliflozin 15 mg (T2DM and With Severe Renal Impairment) | Ertugliflozin 15 mg (Healthy Part. With Normal Renal Function)
Number analyzed (Participants) | 6 | 8 | 8 | 6 | 8
ng•hr/mL | 1559 (21) | 2620 (34) | 3668 (56) | 2742 (41) | 1113 (32)

15. Primary Outcome: Area Under the Plasma Concentration-Time Profile for Glucuronide Metabolite PF-06481944 From Time 0 to the Time of the Last Quantifiable Concentration (AUClast)
Description: Area under the plasma concentration-time profile from Time 0 to the time of the last quantifiable concentration (Clast). Blood samples were taken at pre-dose up to 96 hours post-dose, from which the concentration of glucuronide metabolite PF 06481944 was determined. Geometric Coefficient of Variation was reported as a percent.
Time Frame: Time 0 (predose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, and 96 hours post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng•hr/mL
Arm/Group | Ertugliflozin 15 mg (T2DM With Normal Renal Function) | Ertugliflozin 15 mg (T2DM With Mild Renal Impairment) | Ertugliflozin 15 mg (T2DM With Moderate Renal Impairment) | Ertugliflozin 15 mg (T2DM and With Severe Renal Impairment) | Ertugliflozin 15 mg (Healthy Part. With Normal Renal Function)
Number analyzed (Participants) | 6 | 8 | 8 | 6 | 8
ng•hr/mL | 1536 (21) | 2517 (32) | 3552 (55) | 2642 (40) | 1090 (33)

16. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) for Glucuronide Metabolite PF-06481944
Description: Cmax is a measure of the maximum amount of drug in the plasma after the dose is given. Blood samples were taken at pre-dose up to 96 hours post-dose, from which the concentration of glucuronide metabolite PF 06481944 was determined. Geometric Coefficient of Variation was reported as a percent.
Time Frame: Time 0 (predose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, and 96 hours post-dose
Population: The analysis population was defined as all treated participants who had at least one concentration measurement for Cmax.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Ertugliflozin 15 mg (T2DM With Normal Renal Function) | Ertugliflozin 15 mg (T2DM With Mild Renal Impairment) | Ertugliflozin 15 mg (T2DM With Moderate Renal Impairment) | Ertugliflozin 15 mg (T2DM and With Severe Renal Impairment) | Ertugliflozin 15 mg (Healthy Part. With Normal Renal Function)
Number analyzed (Participants) | 6 | 8 | 8 | 6 | 8
ng/mL | 217.8 (18) | 309.0 (30) | 358.5 (28) | 218.6 (33) | 168.6 (34)

17. Primary Outcome: Time for Cmax (Tmax) for Plasma Glucuronide Metabolite PF-06481944
Description: Tmax is a measure of the time to reach the maximum concentration in the plasma after the drug dose and is observed directly from data as time of first occurrence. Blood samples were taken at pre-dose up to 96 hours post-dose, from which the concentration of glucuronide metabolite PF 06481944 was determined.
Time Frame: Time 0 (predose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, and 96 hours post-dose
Population: The analysis population was defined as all treated participants who had at least one concentration measurement for Tmax.
Measure: Median (Full Range); unit: Hours
Arm/Group | Ertugliflozin 15 mg (T2DM With Normal Renal Function) | Ertugliflozin 15 mg (T2DM With Mild Renal Impairment) | Ertugliflozin 15 mg (T2DM With Moderate Renal Impairment) | Ertugliflozin 15 mg (T2DM and With Severe Renal Impairment) | Ertugliflozin 15 mg (Healthy Part. With Normal Renal Function)
Number analyzed (Participants) | 6 | 8 | 8 | 6 | 8
Hours | 2.00 [1.00 to 3.00] | 2.00 [1.50 to 4.00] | 3.00 [1.50 to 3.00] | 3.00 [1.50 to 4.00] | 2.00 [1.50 to 3.00]

18. Primary Outcome: Terminal Half-life (t1/2) for Plasma Glucuronide Metabolite PF-06481944
Description: T1/2 is the time required for a given drug concentration in the plasma to decrease by 50%. T1/2 = Loge(2)/kel, where kel was the terminal phase rate constant calculated by a linear regression of the log-linear concentration-time curve. Blood samples were taken at pre-dose up to 96 hours post-dose, from which the concentration of glucuronide metabolite PF 06481944 was determined.
Time Frame: Time 0 (predose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, and 96 hours post-dose
Population: The analysis population was defined as all treated participants who had at least one concentration measurement for t1/2.
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Ertugliflozin 15 mg (T2DM With Normal Renal Function) | Ertugliflozin 15 mg (T2DM With Mild Renal Impairment) | Ertugliflozin 15 mg (T2DM With Moderate Renal Impairment) | Ertugliflozin 15 mg (T2DM and With Severe Renal Impairment) | Ertugliflozin 15 mg (Healthy Part. With Normal Renal Function)
Number analyzed (Participants) | 6 | 8 | 8 | 6 | 8
Hours | 16.68 (9.46) | 22.04 (12.15) | 23.33 (6.15) | 22.83 (5.92) | 17.51 (5.69)

19. Primary Outcome: Cumulative Amount of Drug Recovered Unchanged in Urine to 96 Hours Post Dose (Ae96) for Glucuronide Metabolite PF-06481944
Description: as for outcome 9
Time Frame: 0-4, 4-8, 8-12, 12-24, 24-48, 48-72, and 72-96 hours after dosing on Day 1
Population: The analysis population was defined as all treated participants who had at least one concentration measurement for Ae96.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Milligrams
Arm/Group | Ertugliflozin 15 mg (T2DM With Normal Renal Function) | Ertugliflozin 15 mg (T2DM With Mild Renal Impairment) | Ertugliflozin 15 mg (T2DM With Moderate Renal Impairment) | Ertugliflozin 15 mg (T2DM and With Severe Renal Impairment) | Ertugliflozin 15 mg (Healthy Part. With Normal Renal Function)
Number analyzed (Participants) | 6 | 8 | 8 | 6 | 8
Milligrams | 7.056 (32) | 5.861 (36) | 3.768 (40) | 1.630 (41) | 6.225 (32)

20. Primary Outcome: CLr for Urinary Glucuronide Metabolite PF-06481944
Description: as for outcome 11
Time Frame: 0-4, 4-8, 8-12, 12-24, 24-48, 48-72, and 72-96 hours after dosing on Day 1
Population: The analysis population was defined as all treated participants who had at least one concentration measurement for CLr.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/min.
Arm/Group | Ertugliflozin 15 mg (T2DM With Normal Renal Function) | Ertugliflozin 15 mg (T2DM With Mild Renal Impairment) | Ertugliflozin 15 mg (T2DM With Moderate Renal Impairment) | Ertugliflozin 15 mg (T2DM and With Severe Renal Impairment) | Ertugliflozin 15 mg (Healthy Part. With Normal Renal Function)
Number analyzed (Participants) | 6 | 8 | 8 | 6 | 8
mL/min. | 76.28 (24) | 38.73 (58) | 17.67 (56) | 10.27 (80) | 94.53 (25)

21. Primary Outcome: Area Under the Plasma Concentration-Time Profile for Glucuronide Metabolite PF-06685948 From Time 0 Extrapolated to Infinite Time (AUCinf)
Description: Area under the plasma concentration-time profile from Time 0 extrapolated to infinite time. Blood samples were taken at pre-dose up to 96 hours post-dose, from which the concentration of glucuronide metabolite PF-06685948 was determined. Geometric Coefficient of Variation was reported as a percent.
Time Frame: Time 0 (predose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, and 96 hours post-dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng•hr/mL
Arm/Group | Ertugliflozin 15 mg (T2DM With Normal Renal Function) | Ertugliflozin 15 mg (T2DM With Mild Renal Impairment) | Ertugliflozin 15 mg (T2DM With Moderate Renal Impairment) | Ertugliflozin 15 mg (T2DM and With Severe Renal Impairment) | Ertugliflozin 15 mg (Healthy Part. With Normal Renal Function)
Number analyzed (Participants) | 6 | 8 | 8 | 6 | 8
ng•hr/mL | 383.9 (26) | 604.1 (39) | 950.9 (75) | 975.0 (53) | 337.6 (27)

22. Primary Outcome: Area Under the Plasma Concentration-Time Profile for Glucuronide Metabolite PF-06685948 From Time 0 to the Time of the Last Quantifiable Concentration (AUClast)
Description: Area under the plasma concentration-time profile from Time 0 to the time of the last quantifiable concentration (Clast). Blood samples were taken at pre-dose up to 96 hours post-dose, from which the concentration of glucuronide metabolite PF-06685948 was determined. Geometric Coefficient of Variation was reported as a percent.
Time Frame: Time 0 (predose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, and 96 hours post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng•hr/mL
Arm/Group | Ertugliflozin 15 mg (T2DM With Normal Renal Function) | Ertugliflozin 15 mg (T2DM With Mild Renal Impairment) | Ertugliflozin 15 mg (T2DM With Moderate Renal Impairment) | Ertugliflozin 15 mg (T2DM and With Severe Renal Impairment) | Ertugliflozin 15 mg (Healthy Part. With Normal Renal Function)
Number analyzed (Participants) | 6 | 8 | 8 | 6 | 8
ng•hr/mL | 371.9 (27) | 579.8 (37) | 917.7 (74) | 922.1 (51) | 329.1 (28)

23. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) for Glucuronide Metabolite PF-06685948
Description: Cmax is a measure of the maximum amount of drug in the plasma after the dose is given. Blood samples were taken at pre-dose up to 96 hours post-dose, from which the concentration of glucuronide metabolite PF-06685948 was determined. Geometric Coefficient of Variation was reported as a percent.
Time Frame: Time 0 (predose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, and 96 hours post-dose
Population: The analysis population was defined as all treated participants who had at least one concentration measurement for Cmax.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Ertugliflozin 15 mg (T2DM With Normal Renal Function) | Ertugliflozin 15 mg (T2DM With Mild Renal Impairment) | Ertugliflozin 15 mg (T2DM With Moderate Renal Impairment) | Ertugliflozin 15 mg (T2DM and With Severe Renal Impairment) | Ertugliflozin 15 mg (Healthy Part. With Normal Renal Function)
Number analyzed (Participants) | 6 | 8 | 8 | 6 | 8
ng/mL | 44.44 (22) | 53.56 (17) | 63.10 (42) | 46.42 (35) | 43.90 (24)

24. Primary Outcome: Time for Cmax (Tmax) for Plasma Glucuronide Metabolite PF-06685948
Description: Tmax is a measure of the time to reach the maximum concentration in the plasma after the drug dose and is observed directly from data as time of first occurrence. Blood samples were taken at pre-dose up to 96 hours post-dose, from which the concentration of glucuronide metabolite PF-06685948 was determined.
Time Frame: Time 0 (predose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, and 96 hours post-dose
Population: The analysis population was defined as all treated participants who had at least one concentration measurement for Tmax.
Measure: Median (Full Range); unit: Hours
Arm/Group | Ertugliflozin 15 mg (T2DM With Normal Renal Function) | Ertugliflozin 15 mg (T2DM With Mild Renal Impairment) | Ertugliflozin 15 mg (T2DM With Moderate Renal Impairment) | Ertugliflozin 15 mg (T2DM and With Severe Renal Impairment) | Ertugliflozin 15 mg (Healthy Part. With Normal Renal Function)
Number analyzed (Participants) | 6 | 8 | 8 | 6 | 8
Hours | 2.00 [1.50 to 3.00] | 3.00 [2.00 to 4.03] | 4.00 [2.00 to 4.00] | 3.51 [3.00 to 4.02] | 2.00 [2.00 to 3.00]

25. Primary Outcome: Terminal Half-life (t1/2) for Plasma Glucuronide Metabolite PF-06685948
Description: T1/2 is the time required for a given drug concentration in the plasma to decrease by 50%. T1/2 = Loge(2)/kel, where kel was the terminal phase rate constant calculated by a linear regression of the log-linear concentration-time curve. Blood samples were taken at pre-dose up to 96 hours post-dose, from which the concentration of glucuronide metabolite PF-06685948 was determined.
Time Frame: Time 0 (predose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, and 96 hours post-dose
Population: The analysis population was defined as all treated participants who had at least one concentration measurement for t1/2.
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Ertugliflozin 15 mg (T2DM With Normal Renal Function) | Ertugliflozin 15 mg (T2DM With Mild Renal Impairment) | Ertugliflozin 15 mg (T2DM With Moderate Renal Impairment) | Ertugliflozin 15 mg (T2DM and With Severe Renal Impairment) | Ertugliflozin 15 mg (Healthy Part. With Normal Renal Function)
Number analyzed (Participants) | 6 | 8 | 8 | 6 | 8
Hours | 14.87 (7.77) | 21.71 (11.26) | 22.49 (5.30) | 25.22 (10.42) | 15.68 (4.66)

26. Primary Outcome: Cumulative Amount of Drug Recovered Unchanged in Urine to 96 Hours Post Dose (Ae96) for Glucuronide Metabolite PF-06685948
Description: Urine samples were taken at pre-dose up to 96 hours post-dose, from which the concentration of ertugliflozin was determined.
  Ae96 = Sum of [urine concentration × sample volume] for each collection interval from 0 to 96 hours post dose. Blood samples were taken at pre-dose up to 96 hours post-dose, from which the concentration of glucuronide metabolite PF-06685948 was determined. Geometric Coefficient of Variation was reported as a percent.
Time Frame: 0-4, 4-8, 8-12, 12-24, 24-48, 48-72, and 72-96 hours after dosing on Day 1
Population: The analysis population was defined as all treated participants who had at least one concentration measurement for Ae96.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Milligrams
Arm/Group | Ertugliflozin 15 mg (T2DM With Normal Renal Function) | Ertugliflozin 15 mg (T2DM With Mild Renal Impairment) | Ertugliflozin 15 mg (T2DM With Moderate Renal Impairment) | Ertugliflozin 15 mg (T2DM and With Severe Renal Impairment) | Ertugliflozin 15 mg (Healthy Part. With Normal Renal Function)
Number analyzed (Participants) | 6 | 8 | 8 | 6 | 8
Milligrams | 0.9575 (45) | 0.7882 (33) | 0.6603 (49) | 0.3195 (43) | 0.8287 (40)

27. Primary Outcome: Renal Clearance (CLr) for Urinary Glucuronide Metabolite PF-06685948
Description: Urine samples were taken at pre-dose up to 96 hours post-dose, from which the concentration of ertugliflozin was determined.
  CLr is Renal Clearance (Ae96 / AUC96), where Ae96 is the cumulative amount of drug recovered unchanged in urine to 96 hours post dose and AUC96 was the area under the concentration-time profile form time 0 to 96 hours. Blood samples were taken at pre-dose up to 96 hours post-dose, from which the concentration of glucuronide metabolite PF-06685948 was determined. Geometric Coefficient of Variation was reported as a percent.
Time Frame: 0-4, 4-8, 8-12, 12-24, 24-48, 48-72, and 72-96 hours after dosing on Day 1
Population: The analysis population was defined as all treated participants who had at least one concentration measurement for CLr.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/min
Arm/Group | Ertugliflozin 15 mg (T2DM With Normal Renal Function) | Ertugliflozin 15 mg (T2DM With Mild Renal Impairment) | Ertugliflozin 15 mg (T2DM With Moderate Renal Impairment) | Ertugliflozin 15 mg (T2DM and With Severe Renal Impairment) | Ertugliflozin 15 mg (Healthy Part. With Normal Renal Function)
Number analyzed (Participants) | 6 | 8 | 8 | 6 | 8
mL/min | 41.82 (24) | 22.50 (45) | 11.95 (49) | 5.778 (43) | 41.42 (31)

28. Primary Outcome: Change From Baseline in 24 Hour Inhibition of Glucose Reabsorption
Description: Inhibition of Glucose Reabsorption = 100 * urinary glucose excretion / (eGFR(ML/MIN) * Weighted Mean Plasma Glucose * 0.0144). 0.0144 is a unit conversion factor used to make the ratio unitless. Geometric Coefficient of Variation was reported as a percent.
Time Frame: Baseline and 24 Hours
Population: The analysis population was defined as all treated participants who had at least one concentration measurement for plasma glucose concentration.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage
Arm/Group | Ertugliflozin 15 mg (T2DM With Normal Renal Function) | Ertugliflozin 15 mg (T2DM With Mild Renal Impairment) | Ertugliflozin 15 mg (T2DM With Moderate Renal Impairment) | Ertugliflozin 15 mg (T2DM and With Severe Renal Impairment) | Ertugliflozin 15 mg (Healthy Part. With Normal Renal Function)
Number analyzed (Participants) | 6 | 8 | 8 | 6 | 8
Percentage | 33.34 (22) | 25.58 (77) | 28.84 (34) | 24.25 (61) | 29.19 (34)
Statistical Analysis 1: Comparison: Ertugliflozin 15 mg (T2DM With Normal Renal Function) vs Ertugliflozin 15 mg (T2DM With Mild Renal Impairment); Test type: Superiority or Other; Ratio: Mild Ren. Impa./T2DM Norm. Renal = 76.73, 95% CI 2-sided [48.58 to 121.19] — Adjusted geometrics mean values were used. The model was an ANOVA model with renal function group as a fixed effect
Statistical Analysis 2: Comparison: Ertugliflozin 15 mg (T2DM With Normal Renal Function) vs Ertugliflozin 15 mg (T2DM With Moderate Renal Impairment); Test type: Superiority or Other; Ratio: Mod. Ren. Impa./T2DM Norm. Renal = 86.52, 95% CI 2-sided [54.78 to 136.65] — Adjusted geometrics mean values were used. The model was an ANOVA model with renal function group as a fixed effect
Statistical Analysis 3: Comparison: Ertugliflozin 15 mg (T2DM With Normal Renal Function) vs Ertugliflozin 15 mg (T2DM and With Severe Renal Impairment); Test type: Superiority or Other; Ratio: Sev. Ren. Impa./T2DM Norm. Renal = 72.74, 95% CI 2-sided [44.63 to 118.58] — Adjusted geometrics mean values were used. The model was an ANOVA model with renal function group as a fixed effect

29. Primary Outcome: Change From Baseline in 24 Hour Fluid Balance
Description: Fluid balance = fluid intake - urine output.
Time Frame: For 24 hours before Baseline (-48 to -24 hours) and up to 24 hours after dosing on Day 1 (Up to 24 hours)
Population: The analysis population was defined as all treated participants who had at least one measurement for fluid balance.
Measure: Mean (Standard Deviation); unit: Milliliters
Arm/Group | Ertugliflozin 15 mg (T2DM With Normal Renal Function) | Ertugliflozin 15 mg (T2DM With Mild Renal Impairment) | Ertugliflozin 15 mg (T2DM With Moderate Renal Impairment) | Ertugliflozin 15 mg (T2DM and With Severe Renal Impairment) | Ertugliflozin 15 mg (Healthy Part. With Normal Renal Function)
Number analyzed (Participants) | 6 | 8 | 8 | 6 | 8
Milliliters | -660.67 (515.48) [-1132.02 to -189.31] | -937.00 (539.14) [-1345.20 to -528.79] | -696.38 (832.57) [-1104.58 to -288.17] | 111.50 (736.79) [-359.85 to 582.85] | -478.63 (583.02)

30. Secondary Outcome: Urinary Glucose Excretion Over 24 Hours (UGE0-24hr) for Ertugliflozin
Description: Participants were asked to void at the end of each prescribed interval with forced voids prior to start and at the end of each interval.
Time Frame: 0-4, 4-8, 8-12, 12-24 hours after dosing on Day 1
Population: The analysis population was defined as all treated participants who had at least one concentration measurement for UGE0-24hr.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Grams
Arm/Group | Ertugliflozin 15 mg (T2DM With Normal Renal Function) | Ertugliflozin 15 mg (T2DM With Mild Renal Impairment) | Ertugliflozin 15 mg (T2DM With Moderate Renal Impairment) | Ertugliflozin 15 mg (T2DM and With Severe Renal Impairment) | Ertugliflozin 15 mg (Healthy Part. With Normal Renal Function)
Number analyzed (Participants) | 6 | 8 | 8 | 6 | 8
Grams | 72.31 (30) | 35.98 (113) | 27.55 (68) | 10.09 (57) | 46.33 (31)
Statistical Analysis 1: Comparison: Ertugliflozin 15 mg (T2DM With Normal Renal Function) vs Ertugliflozin 15 mg (T2DM With Mild Renal Impairment); Test type: Superiority or Other; Ratio (Mild Renal Impair./T2DM Norm. Ren = 49.75, 90% CI 2-sided [27.22 to 90.93] — The model was an ANOVA model with renal function group as a fixed effect
Statistical Analysis 2: Comparison: Ertugliflozin 15 mg (T2DM With Normal Renal Function) vs Ertugliflozin 15 mg (T2DM With Moderate Renal Impairment); Test type: Superiority or Other; Ratio (Mod. Renal Impair./T2DM Norm. Ren = 38.10, 90% CI 2-sided [20.85 to 69.64] — The model was an ANOVA model with renal function group as a fixed effect
Statistical Analysis 3: Comparison: Ertugliflozin 15 mg (T2DM With Normal Renal Function) vs Ertugliflozin 15 mg (T2DM and With Severe Renal Impairment); Test type: Superiority or Other; Ratio (Sev. Renal Impair./T2DM Norm. Ren = 13.95, 90% CI 2-sided [7.32 to 26.58] — The model was an ANOVA model with renal function group as a fixed effect

ADVERSE EVENTS:
Time Frame: Up to 19 days
Description: An AE is defined as any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease associated with the use of a medical treatment or procedure, regardless of whether it is considered related to the medical treatment or procedure, that occurs during the course of the study.
Groups:
- T2DM Normal Renal Function: Ertugliflozin (15 mg), oral, administered in participants with T2DM and with normal renal function
- T2DM Mild Renal Impairment: Ertugliflozin (15 mg), oral, administered in participants with T2DM and with mild renal impairment
- T2DM Moderate Renal Impairment: Ertugliflozin (15 mg), oral, administered in participants with T2DM and with moderate renal impairment
- T2DM Severe Renal Impairment: Ertugliflozin (15 mg), oral, administered in participants with T2DM and with severe renal impairment
- Healthy Normal Renal Function: Ertugliflozin (15 mg), oral, administered in participants with healthy participants and with normal renal function
Arm/Group | T2DM Normal Renal Function | T2DM Mild Renal Impairment | T2DM Moderate Renal Impairment | T2DM Severe Renal Impairment | Healthy Normal Renal Function
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/8 | 0/8 | 0/6 | 0/8
Other Adverse Events (participants affected / at risk) | 1/6 | 2/8 | 1/8 | 3/6 | 4/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | T2DM Normal Renal Function (N=6) | T2DM Mild Renal Impairment (N=8) | T2DM Moderate Renal Impairment (N=8) | T2DM Severe Renal Impairment (N=6) | Healthy Normal Renal Function (N=8)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Catheter site erythema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vessel puncture site haemorrhage (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Nasal mucosal disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator will provide manuscripts, abstracts, or the full text of any other intended disclosure (poster presentation, invited speaker or guest lecturer presentation, etc.) to the sponsor at least 30 days before they are submitted for publication or otherwise disclosed. If any patent action is required to protect intellectual property rights, investigator agrees to delay the disclosure for a period not to exceed an additional 60 days.